CLINICAL TRIAL: NCT01286090
Title: Double-Blind, Randomized, Placebo-Controlled Trial to Assess Efficacy and Safety of R051619 (Cisapride 10 mg Q.I.D.) Versus Placebo for the Improvement of Symptoms Associated With Exacerbations of Gastroparesis, After Failure of Other Treatments, in Patients With Diabetes Mellitus
Brief Title: An Efficacy and Safety Study of Cisapride for Improving Symptoms Associated With Gastroparesis in Patients With Diabetes Mellitus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Portfolio/CDT Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR003946; CIS-INT-25
Record Dates: First submitted 2011-01-13; First posted 2011-01-31 (Estimated); Last update posted 2011-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: Cisapride (PREPULSID); Placebo; Diabetes mellitus; Diabetic gastroparesis
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Cisapride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): Cisapride One 10-mg tablet taken orally 4 times a day for up to 8 weeks.
  Interventions: Drug: Cisapride
- 002 (Experimental): Placebo One tablet taken orally 4 times a day for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cisapride — One 10-mg tablet taken orally 4 times a day for up to 8 weeks.
  Arms: 001
Drug: Placebo — One tablet taken orally 4 times a day for up to 8 weeks.
  Arms: 002

SUMMARY:
The purpose of this study is to assess the effectiveness of cisapride at improving symptoms associated with gastroparesis (a stomach disorder) in patients with diabetes mellitus.

DETAILED DESCRIPTION:
This is a double-blind (neither the physician nor the patient will know the name of assigned treatment) study to determine the effectiveness of cisapride tablets compared to placebo tablets (a tablet identical in appearance to cisapride but does not contain active drug) at improving symptoms associated with diabetic gastroparesis when administered orally (by mouth) to patients with insulin dependent or non-insulin dependent diabetes mellitus. Gastroparesis is a disorder also called delayed gastric emptying, in which the stomach takes too long to empty food into the small intestine for digestion. Symptoms of gastroparesis may include vomiting, nausea, early feeling of fullness after only a few bites of food, weight loss due to poor absorption of nutrients or low calorie intake, abdominal bloating, poor glycemic (blood sugar) control, lack of appetite, and pain in the stomach area. Patients will take study drug (one 10-mg tablet of cisapride, or one tablet of placebo), orally, 4 times a day, for a period of 8 weeks. Study drug will be taken approximately 15 minutes before each meal and, with a beverage, before going to bed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with insulin dependent or non-insulin dependent diabetes mellitus
* Experienced inadequate responses to, or have been intolerant of, treatment with at least one previous drug therapy for gastroparesis
* Have exacerbation of gastroparesis symptoms requiring medical attention
* Demonstrate delayed gastric emptying as assessed by a [1-13C]-Sodium Acetate Breath Test within 14 days before randomization

Exclusion Criteria:

* Received prior treatment with cisapride
* Have a glycosylated hemoglobin (HbA1c) >10% at screening, as determined by clinical laboratory testing
* Have any upper gastrointestinal (GI) pathology other than diabetic gastroparesis that would require therapy other than that provided in this trial
* Have any organic/neurological disease that is suspected to be causing gastroparesis, other than diabetes
* Currently vomiting, or receiving therapy for a severe exacerbation of gastroparesis, that would prevent the patient from receiving oral therapy or a diet

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2003-07; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in Gastroparesis Cardinal Symptoms Index (GCSI) score | At baseline (Visit 2) and weekly during the treatment phase of the trial for up to 8 weeks

SECONDARY OUTCOMES:
The number of adverse events reported | For the duration of the study (up to 8 weeks)
The type of adverse events reported | For the duration of the study (up to 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.